CLINICAL TRIAL: NCT01855958
Title: Primary Motor Cortex Plasticity and the Bottom up Effect of Deep Intramuscular Needling Stimulation Therapy (DIMST)in Osteoarthritis Chronic Pain
Brief Title: Motor Cortex Plasticity and the Effect of Deep Intramuscular Needling Stimulation Therapy (DIMST) in Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0013
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2015-08

CONDITIONS: Knee Osteoarthritis; Chronic Pain
Keywords: Osteoarthritis; Electro acupuncture; Deep intramuscular stimulation; Transcranial Magnetic Stimulation; Pain pressure threshold; Conditioned pain modulation; Clinical trial
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DIMST (Experimental): The investigators used acupuncture needles with guide tubes (Suzhou Huanqiu Acupuncture Medical Appliance Co. Ltd., 218, China) that were 40 mm in length and 0.25 mm in diameter. The needling in DIMST was applied using an electro acupuncture device (Cosmotron, São Paulo, Brazil) in the dermatomes corresponding to the nerve roots involved in the knee (L1, L2, L3, L4, L5, S1, and S2). DIMST using was administered maintaining a distance from the spinous process line of 2 cm. The anatomic sites of peripheral DIMST were the muscles vastus medialis, rectus femoris, vastus lateralis, tibialis anterior; and the pes anserinus bursae. All subjects received one 30min session using a frequency of 2 Hz.
  Interventions: Procedure: DIMST
- Placebo-sham (Sham Comparator): The investigators used the same electro acupuncture device (Cosmotron, Sao Paulo, Brazil), which was previously set to prevent the current to pass through the electrodes. Subjects were informed that it would be a stimulus of low intensity and high frequency that they probably would not have any sense of it. The electrodes were placed on the same points where the active stimulation was applied while the nerve stimulation unit was left in front of the subject, for 30 minutes. This positioning ensured that the intermittent diode simulating the electrical stimulus was visible and audible.
  Interventions: Procedure: Placebo-sham

INTERVENTIONS:
Procedure: DIMST — The investigators used electro acupuncture of 2 Hz during 30 minutes.
  Other Names: Paraspinal electro acupuncture.
  Arms: DIMST
Procedure: Placebo-sham — Electro acupuncture with rubber electrodes, without current passing.
  Other Names: Electrostimulation with rubber electrodes.
  Arms: Placebo-sham

SUMMARY:
The aim of this study is to evaluate the cortical excitability in pain of knee osteoarthritis (OA), as well as the effect of one session of a kind of electroacupuncture (deep needling intramuscular stimulation therapy - DIMST) in this pain and the cortical excitability after the intervention.

The hypothesis is that cortical excitability is altered in this condition, confirming the findings already described in other chronic pain conditions. The investigators also believe that a session DIMST can reduce pain and alter cortical excitability, restoring its previous activity will occur from chronic pain.

DETAILED DESCRIPTION:
Recent developments in the treatment of chronic pain have shown that the primary motor cortex (M1) is an effective target for neural brain stimulation techniques, such as transcranial magnetic stimulation (TMS). Due to these promising initial results, the plasticity of M1 has also been investigated as a potential marker for chronic pain. TMS studies using single or paired pulse shown changes in M1 plasticity in neuropathic pain and fibromyalgia pain compared to healthy subjects. Thus, there is a decrease in the inhibitory activity of chronic pain that can take a state as shown uninhibited by measuring TMS indexed intracortical inhibition (ICI) and cortical silent period (CSP). Based on these experimental data and clinical studies have been focused on the effects of neuromodulation techniques in M1 excitability. The techniques used to stimulate the peripheral nervous system was investigated using different approaches. The DIMST is a therapy applied to treat peripheral chronic syndromes that may have central components such as myofascial pain. During DIMST, the needles are applied to the spinal segment associated with nerve roots dermatome corresponding to the pathology. This treatment can also be effective in the treatment of diseases that have major peripheral components such as OA. OA is a major cause of suffering and disability in the elderly, having an inflammatory component, such as a factor that contributes to the symptoms and progression of the disease. There is evidence that OA could lead to sensitization central and segmental, but these effects on M1 plasticity and other central components are not completely known.

Therefore, researchers proposed to evaluate the plasticity of M1 in this chronic pain condition and also the effect of bottom-up DIMST in pain and cortical excitability.

ELIGIBILITY:
Inclusion Criteria:

* Women with over 18 years old, with chronic pain because of primary osteoarthritis of the knee.
* Pain stable for at least three months. Score greater than or equal to 3 cm (0 cm = "no pain" and "worst possible pain" = 10cm) on VAS for pain perception at baseline.
* No contraindications to electro acupuncture or transcranial magnetic stimulation.
* Naive in acupuncture treatment.

Exclusion Criteria:

* Clinically significant or unstable disorder, medical or psychiatric.
* Presence of neurological or rheumatic comorbidity.
* Pregnancy.
* Having performed surgery in the knee to be treated in the last 6 months, or be planning surgery for the next semester.
* Having performed with corticosteroid infiltration in the last six weeks or are using this.
* Having performed with hyaluronic acid infiltration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — Federal University of Rio Grande do Sul; Maria L Tarragó, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre., Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Lefaucheur JP, Drouot X, Menard-Lefaucheur I, Keravel Y, Nguyen JP. Motor cortex rTMS restores defective intracortical inhibition in chronic neuropathic pain. Neurology. 2006 Nov 14;67(9):1568-74. doi: 10.1212/01.wnl.0000242731.10074.3c. PMID 17101886
- [Background] Zunhammer M, Eichhammer P, Franz J, Hajak G, Busch V. Effects of acupuncture needle penetration on motor system excitability. Neurophysiol Clin. 2012 Jun;42(4):225-30. doi: 10.1016/j.neucli.2012.02.134. Epub 2012 Mar 6. PMID 22632870
- [Background] Lo YL, Cui SL. Acupuncture and the modulation of cortical excitability. Neuroreport. 2003 Jul 1;14(9):1229-31. doi: 10.1097/00001756-200307010-00008. PMID 12824765
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Schwenkreis P, Scherens A, Ronnau AK, Hoffken O, Tegenthoff M, Maier C. Cortical disinhibition occurs in chronic neuropathic, but not in chronic nociceptive pain. BMC Neurosci. 2010 Jun 11;11:73. doi: 10.1186/1471-2202-11-73. PMID 20540759
- [Background] Laste G, Caumo W, Adachi LN, Rozisky JR, de Macedo IC, Filho PR, Partata WA, Fregni F, Torres IL. After-effects of consecutive sessions of transcranial direct current stimulation (tDCS) in a rat model of chronic inflammation. Exp Brain Res. 2012 Aug;221(1):75-83. doi: 10.1007/s00221-012-3149-x. Epub 2012 Jul 3. PMID 22752510
- [Background] Le Bars D, Dickenson AH, Besson JM. Diffuse noxious inhibitory controls (DNIC). II. Lack of effect on non-convergent neurones, supraspinal involvement and theoretical implications. Pain. 1979 Jun;6(3):305-327. doi: 10.1016/0304-3959(79)90050-2. PMID 460936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a call list generated by public means of mass communication in January 2012, and announcements of research in the Department of Pain and Palliative Medicine, Hospital de Clinicas, before and during the study. Throughout the study the members of the list were selected through a telephone interview.
Pre-assignment Details: Eighty-five subjects were screened. Five refused to participate, fifty-four were not enrolled for the following reasons:
  Previous experience with acupuncture. Inability to walk a certain distance. Live distant of center. Twenty-six were recruited in the study and randomized further to active(n = 13) or placebo (n = 13)groups.
Groups:
- DIMST, Deep Intramuscular Stimulation Therapy: The investigators used acupuncture needles with guide tubes (Suzhou Huanqiu Acupuncture Medical Appliance Co. Ltd., 218, China) that were 40 mm in length and 0.25 mm in diameter. The needling in DIMST was applied using an electro acupuncture device (Cosmotron, São Paulo, Brazil) in the dermatomes corresponding to the nerve roots involved in the knee (L1, L2, L3, L4, L5, S1, and S2). DIMST using was administered maintaining a distance from the spinous process line of 2 cm. The anatomic sites of peripheral DIMST were the muscles vastus medialis, rectus femoris, vastus lateralis, tibialis anterioris; and the pes anserinus bursae. All subjects received one 30min session using a frequency of 2 Hz.
- Placebo-sham, Rubber Electrodes With Electrostimulation: The investigators used the same electro acupuncture device (Cosmotron, Sao Paulo, Brazil), which was previously set to prevent the current to pass through the electrodes. Subjects were informed that it would be a stimulus of low intensity and high frequency that they probably would not have any sense of it. The electrodes were placed on the same points where the active stimulation was applied while the nerve stimulation unit was left in front of the subject, for 30 minutes. This positioning ensured that the intermittent diode simulating the electrical stimulus was visible and audible.
Period: Overall Study
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.85 (7.53) | 63.55 (7.54) | 64.50 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 13 | 13 | 26

OUTCOME MEASURES:

1. Secondary Outcome: Intracortical Inhibition (ICI) After Intervention.
Description: ICI was evaluated using inter-stimuli intervals (ISIs) of 2 ms with paired-pulse stimulation. The subthreshold stimulus was set at 80% of rMT (conditioning stimulus) , and the suprathreshold test stimulus was set at 130% of rMT. After a randomized protocol, thirty stimuli were assessed using a 2ms interval (ICI), a 12ms interval (ICF) and test-only trials (MEPs). The resulting MEP amplitude was converted into the mean amplitude, and paired-pulse parameters were expressed as the amount of inhibition or facilitation. The calculation result of ICI was done by the ratio of the mean ICI by the mean MEP.
  # Below the data after intervention.
Time Frame: Evaluated in one day. The cortical excitability before and within an hour after intervention.
Measure: Mean (Standard Deviation); unit: ratio of amplitude (mV).
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Number analyzed (Participants) | 13 | 13
ratio of amplitude (mV). | 0.75 (0.72) | 0.57 (0.30)

2. Secondary Outcome: Pain Intensity After Intervention.
Description: The intensity of pain was measured by a 10-cm VAS. VAS scores ranged from no pain (zero) to the worst possible pain possible (10 cm). The pain score on VAS during the last 24 hours was used to classify the subjects into two groups: (1) absence of pain or mild pain (scores equal to or lower than 4 cm) and (2) moderate, intense, or worst possible pain (scores higher than 4 cm).
  # Below the data after intervention.
Time Frame: Evaluated within twenty four hours before and within one hour after the intervention.
Measure: Mean (Standard Deviation); unit: cm ( mean).
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Number analyzed (Participants) | 13 | 13
cm ( mean). | 0.88 (1.58) | 3.36 (3.32)

3. Primary Outcome: Pain Pressure Threshold (PPT) After Intervention..
Description: PPT (alone): The patient was instructed to verbally report the perception of pain onset. The investigator assessed PPT using an electronic algometer (J Tech Medical Industries, USA). The device had a 1-cm2 hard-rubber probe, which was applied over structures at L1- L5 dermatome at the knee and at the contralateral forearm. The average values of PPT in kgf/cm2 for three successive readings taken at intervals of 3-5 min were used as the outcomes.
  # Below, the data after intervention.
Time Frame: Before and within one hour after intervention.
Measure: Mean (Standard Deviation); unit: Kgf / cm2
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Number analyzed (Participants) | 13 | 13
Kgf / cm2 | 8.82 (3.00) | 6.66 (1.67)

4. Primary Outcome: Motor Evoked Potential (MEP) After Intervention.
Description: Cortical excitability was assessed using a MagPro X100 (MagVenture Company, Lucernemarken, Denmark) and a figure-of-8 coil centered over the left motor cortex (M1). Subjects were seated in a comfortable reclining chair with their arms and hands lying relaxed on the armrests. The investigators measured the resting motor threshold (rMT) of the right first dorsal interosseous (FDI) muscle. The MEPs were recorded by surface electromyography (EMG) using Ag-AgCl cup electrodes in a belly tendon montage. Resting motor threshold (rMT) was deﬁned as the stimulus intensity at which peak-to-peak MEP amplitude of 50 µV (microvolts) was obtained in at least 5 of 10 consecutive trials.
  MEP was deﬁned as approximately 130% of the rMT or the stimulus intensity at which peak-to-peak MEP amplitude of at least 1 mV was obtained in 10 consecutive trials. The result of the MEP was the average of 10 curves (unconditioned MEP).
  # Below the data after intervention.
Time Frame: Before and within one hour after intervention.
Measure: Mean (Standard Deviation); unit: mV (millivolts).
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Number analyzed (Participants) | 13 | 13
mV (millivolts). | 1.14 (0.83) | 1.12 (1.00)

5. Secondary Outcome: Intracortical Facilitation (ICF) After Intervention.
Description: ICF was evaluated using an inter-stimuli intervals (ISIs) of 12 ms with paired-pulse and similar parameters for the conditioning and test stimuli. After a randomized protocol, thirty stimuli were assessed using a 2ms interval (ICI), a 12ms interval (ICF) and test-only trials (MEP). The resulting MEP amplitude was converted into the mean amplitude, and paired-pulse parameters were expressed as the amount of inhibition or facilitation. The calculation result of ICF was done by the ratio of the mean ICF by the mean MEP.
  # Below the data after intervention.
Time Frame: Before and within one hour after intervention.
Measure: Mean (Standard Deviation); unit: ratio of amplitude (mV).
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Number analyzed (Participants) | 13 | 13
ratio of amplitude (mV). | 1.20 (0.98) | 0.78 (0.57)

6. Secondary Outcome: Cortical Silent Period (CSP) After Intervention.
Description: To determine the cortical silent period (CSP), subjects were instructed to squeeze the dynamometer using their fingers at 20% of maximal force when a single pulse stimulus (130% rMT) was applied. The result was the average of five consecutive measurements. The CSP was determined by the interval between the stimulus and the motor response elicited in the subject.
  # Below the data after intervention.
Time Frame: Evaluated before and within one hour after intervention.
Measure: Mean (Standard Deviation); unit: ms (milliseconds).
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Number analyzed (Participants) | 13 | 13
ms (milliseconds). | 50.93 (24.48) | 48.92 (22.82)

7. Primary Outcome: Conditioned Pain Modulation (CPM) After Intervention.
Description: PPT during cold water immersion (PPT+CPM): By measuring PPT during cold water immersion, we evaluated the degree to which pain perception is modulated by conditioned pain modulation (CPM) following the presentation of an initial heterotopic noxious stimulus. Subjects immersed their left hands into cold water (zero to 1°C) for 1 minute. During the last 30 seconds of cold-water immersion, the PPT procedure was administered at the right forearm. The temperature was held constant across during the experiment for each subject.
  # Below the data after intervention.
Time Frame: Before and within one hour after intervention.
Measure: Mean (Standard Deviation); unit: Kgf / cm2
Arm/Group | DIMST | Placebo-sham
Number analyzed (Participants) | 13 | 13
Kgf / cm2 | 12.62 (3.47) | 9.15 (2.17)

ADVERSE EVENTS:
Arm/Group | DIMST, Deep Intramuscular Stimulation Therapy | Placebo-sham, Rubber Electrodes With Electrostimulation
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No